CLINICAL TRIAL: NCT04708639
Title: Monitoring Alectinib Treatment by Detection of ALK Translocations in Serial Blood Samples From Non-Small Cell Lung Cancer Patients
Acronym: MonAlec
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Aarhus University Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Peter Meldgaard, MD PhD, Aarhus University Hospital
Other Study IDs: ML40920
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer; ALK Gene Mutation; Resistance, Disease; Mutation
MeSH Terms: conditions — Lung Neoplasms; Disease Resistance | interventions — alectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA from blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Alectinib — Use of ctDNA to establish response and resistance to alectinib.

SUMMARY:
Circulating tumor DNA can be used to monitor the treatment effect and identify developing resistance mutations during ALK directed TKI treatment.

DETAILED DESCRIPTION:
The purpose and objectives of the non-interventional study with primary data collection is

* To determine if monitoring the amount of translocated DNA in the blood reflects alectinib treatment effect.
* To assess the presence and type of resistance mutations using ctDNA at the time patients experience clinical progression on alectinib.
* To investigate if the resistance mutations identified at clinical progression could have been identified in blood samples taken before clinically evident progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ALK translocated metastatic NSCLC, treated with alectinib as 1st line therapy in routine clinical practice
2. Written (personally dated and signed) informed consent

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All newly diagnosed ALK translocated lung cancer adenocarcinomas.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS on alectinib | 46 month
  time from initiation of treatment to progression
mechanism of resistance | 15.2 month
  ctDNA to establish resistance mechanisms to alectinib treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Meldgaard, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
All data will be published